CLINICAL TRIAL: NCT01933672
Title: A Phase 1b, Randomized, Double-blind, Active Comparator Controlled, 3-period, Cross-over Study To Characterize The Pharmacodynamics And Tolerability Of Two Dosing Regimens Of Pf-04937319 In Adults With Type 2 Diabetes Mellitus Inadequately Controlled On Metformin
Brief Title: Study Of Two Dosing Regimens Of PF-04937319 Compared To An Approved Agent (Sitagliptin) In Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: B1621019
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Results first posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Phase 1b; type 2 diabetes; metformin background; PF-04937319
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF-04937319 once-daily (Experimental)
  Interventions: Drug: PF-04937319 once-daily
- PF-04937319 split-dose (Experimental)
  Interventions: Drug: PF-04937319 split-dose
- Sitagliptin once-daily (Active Comparator)
  Interventions: Drug: Sitagliptin once-daily

INTERVENTIONS:
Drug: PF-04937319 once-daily — Tablets, 300 mg once-daily with breakfast, 14-days
  Arms: PF-04937319 once-daily
Drug: PF-04937319 split-dose — tablets, 150 mg with breakfast plus 100 mg with lunch, 14-days
  Arms: PF-04937319 split-dose
Drug: Sitagliptin once-daily — tablets, 100 mg once-daily with breakfast, 14-days
  Arms: Sitagliptin once-daily

SUMMARY:
Study B1621019 will assess efficacy and safety of two different dosing regimens of an investigational agent (PF-04937319) compared to an approved drug (sitagliptin) in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes, on background metformin therapy either alone or with 1 other oral anti-diabetic agent (excluding Actos)

Exclusion Criteria:

* Patients with cardiovascular event within 6-months of screening
* Patients with diabetic complications
* Female subjects who are pregnant or planning to become pregnant
* Subjects with unstable medical conditions (eg, hypertension)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - Avail Clinical Research, LLC, DeLand, Florida
  - Miami Research Associates, Inc., South Miami, Florida
  - MRA Clinical Research, LLC, South Miami, Florida
  - High Point Clinical Trials Center, LLC, High Point, North Carolina
  - Community Research, Cincinnati, Ohio
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas
  - Spaulding Clinical Research, LLC, West Bend, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1621019&StudyName=Study%20Of%20Two%20Dosing%20Regimens%20Of%20PF-04937319%20Compared%20To%20An%20Approved%20Agent%20%28Sitagliptin%29%20In%20Patients%20With%20Type%202%20Diabetes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 90 participants with type 2 diabetes mellitus (T2DM) consented for this study; of these, 47 participants were ineligible at screening visit, 43 (47.8%) transitioned into run-in phase where participants were standardized on Sponsor-provided metformin.
Pre-assignment Details: A total of 33 (33/90; 36.7%) participants completed metformin run-in period and were randomized and received to at least one regimen (PF-04937319 split-dose, PF-04937319 once daily, or sitagliptin).
Groups:
- Metformin Run-in: Sponsor-provided, open-label metformin was administered from the run-in visit to the follow-up visit, inclusive, and it was provided as 500 milligram (mg) immediate-release tablets.
- PF-04937319 150+100mg Then PF-04937319 300mg Then Sitagliptin: Participants received the morning dose of PF-04937319 150 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day and the second dose (PF-04937319 100mg) was taken with the lunch meal 5±1 hours after the morning dose, each day, for 14±2 days in the first intervention period; and then received the morning dose of PF-04937319 300 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day, and the second dose of the study medication (placebo) was taken with the lunch meal 5±1 hours after the morning dose each day for 14±2 days in the second intervention period; and then received the morning dose of sitagliptin 100 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day, and the second dose of the study medication (placebo) was taken with the lunch meal 5±1 hours after the morning dose each day for 14±2 days in the third intervention period.
- PF-04937319 150+100mg Then Sitagliptin Then PF-04937319 300mg: Participants received the morning dose of PF-04937319 150 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day and the second dose (PF-04937319 100mg) was taken with the lunch meal 5±1 hours after the morning dose, each day, for 14±2 days in the first intervention period; and then received the morning dose of sitagliptin 100 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day, and the second dose of the study medication (placebo) was taken with the lunch meal 5±1 hours after the morning dose each day for 14±2 days in the second intervention period; and then received the morning dose of PF-04937319 300 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day, and the second dose of the study medication (placebo) was taken with the lunch meal 5±1 hours after the morning dose each day for 14±2 days in the third intervention period.
- PF-04937319 300mg Then PF-04937319 150+100mg Then Sitagliptin: Participants received the morning dose of PF-04937319 300 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day, and the second dose of the study medication (placebo) was taken with the lunch meal 5±1 hours after the morning dose each day for 14±2 days in the first intervention period; and then received the morning dose of PF-04937319 150 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day and the second dose (PF-04937319 100mg) was taken with the lunch meal 5±1 hours after the morning dose, each day, for 14±2 days in the second intervention period; and then received the morning dose of sitagliptin 100 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day, and the second dose of the study medication (placebo) was taken with the lunch meal 5±1 hours after the morning dose each day for 14±2 days.
- PF-04937319 300mg Then Sitagliptin Then PF-04937319 150+100mg: Participants received the morning dose of PF-04937319 300 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day, and the second dose of the study medication (placebo) was taken with the lunch meal 5±1 hours after the morning dose each day for 14±2 days in the first intervention period; and then received the morning dose of sitagliptin 100 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day, and the second dose of the study medication (placebo) was taken with the lunch meal 5±1 hours after the morning dose each day for 14±2 days in the second intervention period; and then received the morning dose of PF-04937319 150 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day and the second dose (PF-04937319 100mg) was taken with the lunch meal 5±1 hours after the morning dose, each day, for 14±2 days in the first intervention period.
- Sitagliptin Then PF-04937319 150+100mg Then PF-04937319 300mg: Participants received the morning dose of sitagliptin 100 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day, and the second dose of the study medication (placebo) was taken with the lunch meal 5±1 hours after the morning dose each day for 14±2 days in the first intervention period; and then received the morning dose of PF-04937319 150 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day and the second dose (PF-04937319 100mg) was taken with the lunch meal 5±1 hours after the morning dose, each day, for 14±2 days in the second intervention period; and then received the morning dose of PF-04937319 300 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day, and the second dose of the study medication (placebo) was taken with the lunch meal 5±1 hours after the morning dose each day for 14±2 days in the third intervention period.
- Sitagliptin Then PF-04937319 300mg Then PF-04937319 150+100mg: Participants received the morning dose of sitagliptin 100 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day, and the second dose of the study medication (placebo) was taken with the lunch meal 5±1 hours after the morning dose each day for 14±2 days in the first intervention period; and then received the morning dose of PF-04937319 300 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day, and the second dose of the study medication (placebo) was taken with the lunch meal 5±1 hours after the morning dose each day for 14±2 days in the second intervention period; and then received the morning dose of PF-04937319 150 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day and the second dose (PF-04937319 100mg) was taken with the lunch meal 5±1 hours after the morning dose, each day, for 14±2 days in the third intervention period.
Period: Metformin Run-in Period
Arm/Group | Metformin Run-in | PF-04937319 150+100mg Then PF-04937319 300mg Then Sitagliptin | PF-04937319 150+100mg Then Sitagliptin Then PF-04937319 300mg | PF-04937319 300mg Then PF-04937319 150+100mg Then Sitagliptin | PF-04937319 300mg Then Sitagliptin Then PF-04937319 150+100mg | Sitagliptin Then PF-04937319 150+100mg Then PF-04937319 300mg | Sitagliptin Then PF-04937319 300mg Then PF-04937319 150+100mg
Started | 43 | 0 | 0 | 0 | 0 | 0 | 0
Received Treatment | 43 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 33 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No longer meets eligibility criteria | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 5 | 0 | 0 | 0 | 0 | 0 | 0
Period: First Intervention Period (12-16 Days)
Arm/Group | Metformin Run-in | PF-04937319 150+100mg Then PF-04937319 300mg Then Sitagliptin | PF-04937319 150+100mg Then Sitagliptin Then PF-04937319 300mg | PF-04937319 300mg Then PF-04937319 150+100mg Then Sitagliptin | PF-04937319 300mg Then Sitagliptin Then PF-04937319 150+100mg | Sitagliptin Then PF-04937319 150+100mg Then PF-04937319 300mg | Sitagliptin Then PF-04937319 300mg Then PF-04937319 150+100mg
Started | 0 | 7 | 3 | 5 | 7 | 5 | 6
Completed | 0 | 7 | 2 | 5 | 6 | 4 | 6
Not Completed | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 1 | 0
Period: First Washout Period (7-14 Days)
Arm/Group | Metformin Run-in | PF-04937319 150+100mg Then PF-04937319 300mg Then Sitagliptin | PF-04937319 150+100mg Then Sitagliptin Then PF-04937319 300mg | PF-04937319 300mg Then PF-04937319 150+100mg Then Sitagliptin | PF-04937319 300mg Then Sitagliptin Then PF-04937319 150+100mg | Sitagliptin Then PF-04937319 150+100mg Then PF-04937319 300mg | Sitagliptin Then PF-04937319 300mg Then PF-04937319 150+100mg
Started | 0 | 7 | 2 | 5 | 6 | 4 | 6
Completed | 0 | 7 | 2 | 5 | 6 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention Period (12-16 Days)
Arm/Group | Metformin Run-in | PF-04937319 150+100mg Then PF-04937319 300mg Then Sitagliptin | PF-04937319 150+100mg Then Sitagliptin Then PF-04937319 300mg | PF-04937319 300mg Then PF-04937319 150+100mg Then Sitagliptin | PF-04937319 300mg Then Sitagliptin Then PF-04937319 150+100mg | Sitagliptin Then PF-04937319 150+100mg Then PF-04937319 300mg | Sitagliptin Then PF-04937319 300mg Then PF-04937319 150+100mg
Started | 0 | 7 | 2 | 5 | 6 | 4 | 6
Completed | 0 | 6 | 1 | 5 | 6 | 4 | 6
Not Completed | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 1 | 0 | 0 | 0 | 0
Period: Second Washout Period (7-14 Days)
Arm/Group | Metformin Run-in | PF-04937319 150+100mg Then PF-04937319 300mg Then Sitagliptin | PF-04937319 150+100mg Then Sitagliptin Then PF-04937319 300mg | PF-04937319 300mg Then PF-04937319 150+100mg Then Sitagliptin | PF-04937319 300mg Then Sitagliptin Then PF-04937319 150+100mg | Sitagliptin Then PF-04937319 150+100mg Then PF-04937319 300mg | Sitagliptin Then PF-04937319 300mg Then PF-04937319 150+100mg
Started | 0 | 6 | 1 | 5 | 6 | 4 | 6
Completed | 0 | 6 | 1 | 5 | 6 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention Period (12-16 Days)
Arm/Group | Metformin Run-in | PF-04937319 150+100mg Then PF-04937319 300mg Then Sitagliptin | PF-04937319 150+100mg Then Sitagliptin Then PF-04937319 300mg | PF-04937319 300mg Then PF-04937319 150+100mg Then Sitagliptin | PF-04937319 300mg Then Sitagliptin Then PF-04937319 150+100mg | Sitagliptin Then PF-04937319 150+100mg Then PF-04937319 300mg | Sitagliptin Then PF-04937319 300mg Then PF-04937319 150+100mg
Started | 0 | 6 | 1 | 5 | 6 | 4 | 6
Completed | 0 | 5 | 1 | 4 | 6 | 4 | 6
Not Completed | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomized to 1 of the 6 treatment sequences (ABC, ACB, BAC, BCA, CAB, and CBA) of PF split dose (150+100 mg) (Treatment A), PF once daily (300 mg) (Treatment B) and sitagliptin 100 mg QD (Treatment C).
Groups:
- All*: A total of 90 participants with T2DM were consented for this study; of these, 43 transitioned into run-in with Sponsor-provided metformin and a total of 33 participants were randomized.
Arm/Group | All*
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weighted Mean Daily Glucose (WMDG) at Day 14
Description: Plasma glucose concentration was determined predose (Hour 0) and at 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 16, 20, and 24 hours postdose on Days 0 (baseline) and 14. WMDG was calculated as the area under the curve (AUC) of the 12-point plasma glucose concentration-time profile divided by 24 hours.
Time Frame: Prior to morning dose (Hour 0) and at 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 16, 20, and 24 hours post morning dose on Days 0 (baseline) and Day 14
Population: Full analysis set defined as all randomized subjects who had taken at least 1 dose of blinded study medication and who had both a baseline and a post-baseline WMDG assessment. Number of participants analyzed was the evaluable participants with a measurement at both baseline and on Day 14.
Measure: Least Squares Mean (Standard Error); unit: milligram/deciliter (mg/dL)
Groups:
- PF-04937319 Split-Dose (150+100 mg): Participants were instructed to take the morning dose of PF-04937319 150 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day. In addition, the second dose of the study medication (PF-04937319 100 mg) should have been taken with the lunch meal approximately 5±1 hours after the morning dose, each day, for 14±2 days.
- PF-04937319 Once-Daily (300 mg): Participants were instructed to take the morning dose of PF-04937319 300 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day. In addition, the second dose of the study medication (placebo) should have been taken with the lunch meal approximately 5±1 hours after the morning dose, each day, for 14±2 days.
- Sitagliptin 100 mg: Participants were instructed to take the morning dose of Sitagliptin 100 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day. In addition, the second dose of the study medication ()placebo should have been taken with the lunch meal approximately 5±1 hours after the morning dose, each day, for 14±2 days.
Arm/Group | PF-04937319 Split-Dose (150+100 mg) | PF-04937319 Once-Daily (300 mg) | Sitagliptin 100 mg
Number analyzed (Participants) | 29 | 30 | 25
milligram/deciliter (mg/dL) | -31.24 (3.952) [NA to NA] | -31.33 (4.604) [NA to NA] | -19.24 (4.437) [NA to NA]
Statistical Analysis 1: Comparison: PF-04937319 Split-Dose (150+100 mg); Change from baseline; Test type: Superiority or Other; Mean Difference (Final Values) = -31.24, 80% CI 2-sided [-36.35 to -26.12]
Statistical Analysis 2: Comparison: PF-04937319 Once-Daily (300 mg); Change from baseline; Test type: Superiority or Other; Median Difference (Final Values) = -31.33, 80% CI 2-sided [-37.29 to -25.37]
Statistical Analysis 3: Comparison: Sitagliptin 100 mg; Change from baseline; Test type: Superiority or Other; Mean Difference (Final Values) = -19.24, 80% CI 2-sided [-24.99 to -13.50]
Statistical Analysis 4: Comparison: PF-04937319 Split-Dose (150+100 mg) vs Sitagliptin 100 mg; There was no hypothesis to be tested. Difference in change from baseline in WMDG between the 2 treatment groups was calculated based on the mixed effects repeated measures model; Test type: Superiority or Other; Mean Difference (Final Values) = -11.99, 80% CI 2-sided [-19.81 to -4.17]
Statistical Analysis 5: Comparison: PF-04937319 Once-Daily (300 mg) vs Sitagliptin 100 mg; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; Mean Difference (Final Values) = -12.09, 80% CI 2-sided [-19.81 to -4.17]

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Day 14
Description: Blood samples for measurement of glucose to permit derivation of pre-meal collections at the pre-specified nominal timepoints of each period: predose (ie, time "0"), 1.5, 3, 5, 6.5, 8, 11, 12.5, 14, 16 and 20 hours on Day 0 (baseline) and Day 14; and predose on Days 1 and 15.
Time Frame: Day 14
Population: Full analysis set defined as all randomized subjects who had taken at least 1 dose of blinded study medication and who had both a baseline and a post-baseline WMDG assessment. Number of participants analyzed was the evaluable participants with a measurement on Day 14.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | PF-04937319 Split-Dose (150+100 mg) | PF-04937319 Once-Daily (300 mg) | Sitagliptin 100 mg
Number analyzed (Participants) | 31 | 30 | 26
mg/dL | -21.92 (3.909) | -20.70 (4.324) | -16.51 (4.419)
Statistical Analysis 1: Comparison: PF-04937319 Split-Dose (150+100 mg); Compared with Baseline; Test type: Superiority or Other; Mean Difference (Final Values) = -21.92, 80% CI 2-sided [-27.00 to -16.85]
Statistical Analysis 2: Comparison: PF-04937319 Once-Daily (300 mg); Compared with Baseline; Test type: Superiority or Other; Mean Difference (Final Values) = -20.70, 80% CI 2-sided [-26.30 to -15.10]
Statistical Analysis 3: Comparison: Sitagliptin 100 mg; Compared with Baseline; Test type: Superiority or Other; Mean Difference (Final Values) = -16.51, 80% CI 2-sided [-22.24 to -10.78]
Statistical Analysis 4: Comparison: PF-04937319 Split-Dose (150+100 mg) vs Sitagliptin 100 mg; Change from baseline in FPG was analyzed in a mixed model analysis of covariance (ANCOVA) with regimen, period, sequence, treatment × period, and carryover as fixed effects. Subjects within sequences were modelled as random effects, with each subject's period-specific baseline response included, as fixed covariates; Test type: Superiority or Other; Median Difference (Final Values) = -5.41, 80% CI 2-sided [-11.74 to 0.92]
Statistical Analysis 5: Comparison: PF-04937319 Once-Daily (300 mg) vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; Mean Difference (Final Values) = -4.19, 80% CI 2-sided [-10.86 to 2.49]

3. Secondary Outcome: Change From Baseline in Pre-meal C-Peptide on Day 14
Description: Blood samples for measurement of glucose to permit derivation of pre-meal collections of blood samples for C-peptide at the pre-specified nominal timepoints at predose, 5 and 11 hours on Day 0 (baseline) and Day 14.
Time Frame: Day 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nanograms/milliliter (ng/mL)
Arm/Group | PF-04937319 Split-Dose (150+100 mg) | PF-04937319 Once-Daily (300 mg) | Sitagliptin 100 mg
Number analyzed (Participants) | 31 | 30 | 26
nanograms/milliliter (ng/mL)
  Pre-breakfast change from baseline | -0.06 (0.101) | 0.06 (0.115) | 0.30 (0.112)
  Pre-lunch change from baseline | 0.20 (0.218) | 0.70 (0.249) | 0.06 (0.242)
  Pre-dinner change from baseline | 0.36 (0.251) | 0.30 (0.289) | 0.32 (0.280)
Statistical Analysis 1: Comparison: PF-04937319 Split-Dose (150+100 mg); Compared with Baseline （Pre-breakfast）; Test type: Superiority or Other; Mean Difference (Final Values) = -0.06, 80% CI 2-sided [-0.19 to 0.07]
Statistical Analysis 2: Comparison: PF-04937319 Once-Daily (300 mg); Compared with Baseline (Pre-breakfast); Test type: Superiority or Other; Mean Difference (Final Values) = 0.06, 80% CI 2-sided [-0.09 to 0.21]
Statistical Analysis 3: Comparison: Sitagliptin 100 mg; Compared with Baseline (Pre-breakfast); Test type: Superiority or Other; Mean Difference (Final Values) = 0.30, 80% CI 2-sided [0.16 to 0.45]
Statistical Analysis 4: Comparison: PF-04937319 Split-Dose (150+100 mg) vs Sitagliptin 100 mg; Pre-breakfast; Time-matched change from baseline in pre-meal C-peptide on Day 14 was analyzed using a mixed effects model with sequence, period, treatment, the treatment by-time interaction, period-specific baseline and carryover as fixed effects. Subjects within sequences were modeled as random effects; Test type: Superiority or Other; Mean Difference (Final Values) = -0.36, 80% CI 2-sided [-0.56 to -0.36]
Statistical Analysis 5: Comparison: PF-04937319 Once-Daily (300 mg) vs Sitagliptin 100 mg; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.24, 80% CI 2-sided [-0.45 to -0.03]
Statistical Analysis 6: Comparison: PF-04937319 Split-Dose (150+100 mg); Compared with Baseline (Pre-lunch); Test type: Superiority or Other; Mean Difference (Final Values) = 0.20, 80% CI 2-sided [-0.08 to 0.48]
Statistical Analysis 7: Comparison: PF-04937319 Once-Daily (300 mg); Compared with Baseline (Pre-lunch); Test type: Superiority or Other; Mean Difference (Final Values) = 0.70, 80% CI 2-sided [0.38 to 1.03]
Statistical Analysis 8: Comparison: Sitagliptin 100 mg; Compared with Baseline (Pre-lunch); Test type: Superiority or Other; Mean Difference (Final Values) = 0.06, 80% CI 2-sided [-0.26 to 0.37]
Statistical Analysis 9: Comparison: PF-04937319 Split-Dose (150+100 mg) vs Sitagliptin 100 mg; Pre-lunch; Time-matched change from baseline in pre-meal C-peptide on Day 14 was analyzed using a mixed effects model with sequence, period, treatment, the treatment by-time interaction, period-specific baseline and carryover as fixed effects. Subjects within sequences were modeled as random effects; Test type: Superiority or Other; Mean Difference (Final Values) = 0.14, 80% CI [-0.28 to 0.57]
Statistical Analysis 10: Comparison: PF-04937319 Once-Daily (300 mg) vs Sitagliptin 100 mg; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.65, 80% CI 2-sided [0.19 to 1.11]
Statistical Analysis 11: Comparison: PF-04937319 Split-Dose (150+100 mg); Compared with Baseline (Pre-dinner); Test type: Superiority or Other; Mean Difference (Final Values) = 0.36, 80% CI 2-sided [0.03 to 0.68]
Statistical Analysis 12: Comparison: PF-04937319 Once-Daily (300 mg); Compared with Baseline (Pre-dinner); Test type: Superiority or Other; Mean Difference (Final Values) = 0.30, 80% CI 2-sided [-0.08 to 0.67]
Statistical Analysis 13: Comparison: Sitagliptin 100 mg; Compared with Baseline (Pre-dinner); Test type: Superiority or Other; Mean Difference (Final Values) = 0.32, 80% CI 2-sided [-0.05 to 0.68]
Statistical Analysis 14: Comparison: PF-04937319 Split-Dose (150+100 mg) vs Sitagliptin 100 mg; Pre-dinner; Time-matched change from baseline in pre-meal C-peptide on Day 14 was analyzed using a mixed effects model with sequence, period, treatment, the treatment by-time interaction, period-specific baseline and carryover as fixed effects. Subjects within sequences were modeled as random effects; Test type: Superiority or Other; Mean Difference (Final Values) = 0.04, 80% CI 2-sided [-0.45 to 0.53]
Statistical Analysis 15: Comparison: PF-04937319 Once-Daily (300 mg) vs Sitagliptin 100 mg; [analysis description as in outcome 3, analysis 14]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.02, 80% CI 2-sided [-0.55 to 0.51]

4. Secondary Outcome: Change From Baseline in Pre-meal Insulin on Day 14
Description: Blood samples for measurement of glucose to permit derivation of pre-meal collections of blood samples for insulin at 0, 5 and 11 hours on Day 0 (baseline) and Day 14.
Time Frame: Day 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: micro international unit/milliliter
Arm/Group | PF-04937319 Split-Dose (150+100 mg) | PF-04937319 Once-Daily (300 mg) | Sitagliptin 100 mg
Number analyzed (Participants) | 31 | 30 | 26
micro international unit/milliliter
  Pre-breakfast (n=31,30,26) | 0.16 (0.704) | 0.46 (0.810) | 1.60 (0.793)
  Pre-lunch (n=30,27,25) | 1.69 (1.690) | 4.07 (1.939) | -0.01 (1.864)
  Pre-dinner (n=30,28,24) | -0.70 (2.286) | 5.06 (2.597) | 3.42 (2.714)
Statistical Analysis 1: Comparison: PF-04937319 Split-Dose (150+100 mg); Compared with Baseline （Pre-breakfast）; Test type: Superiority or Other; Mean Difference (Final Values) = 0.16, 80% CI 2-sided [-0.75 to 1.07]
Statistical Analysis 2: Comparison: PF-04937319 Once-Daily (300 mg); Compared with Baseline (Pre-breakfast); Test type: Superiority or Other; Mean Difference (Final Values) = 0.46, 80% CI 2-sided [-0.58 to 1.51]
Statistical Analysis 3: Comparison: Sitagliptin 100 mg; Compared with Baseline (Pre-breakfast); Test type: Superiority or Other; Mean Difference (Final Values) = 1.60, 80% CI 2-sided [0.58 to 2.63]
Statistical Analysis 4: Comparison: PF-04937319 Split-Dose (150+100 mg) vs Sitagliptin 100 mg; Pre-breakfast; Time-matched change from baseline in pre-meal insulin on Day 14 was analyzed using a mixed effects model with sequence, period, treatment, the treatment by-time interaction, period-specific baseline and carryover as fixed effects. Subjects within sequences were modeled as random effects; Test type: Superiority or Other; Mean Difference (Final Values) = -1.45, 80% CI 2-sided [-2.84 to -0.05]
Statistical Analysis 5: Comparison: PF-04937319 Once-Daily (300 mg) vs Sitagliptin 100 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; Median Difference (Final Values) = -1.14, 80% CI 2-sided [-2.63 to 0.35]
Statistical Analysis 6: Comparison: PF-04937319 Split-Dose (150+100 mg); Compared with Baseline (Pre-lunch); Test type: Superiority or Other; Mean Difference (Final Values) = 1.69, 80% CI 2-sided [-0.50 to 3.88]
Statistical Analysis 7: Comparison: PF-04937319 Once-Daily (300 mg); Compared with Baseline (Pre-lunch); Test type: Superiority or Other; Mean Difference (Final Values) = 4.07, 80% CI 2-sided [1.56 to 6.58]
Statistical Analysis 8: Comparison: Sitagliptin 100 mg; Compared with Baseline (Pre-lunch); Test type: Superiority or Other; Mean Difference (Final Values) = -0.01, 80% CI 2-sided [-2.42 to 2.40]
Statistical Analysis 9: Comparison: PF-04937319 Split-Dose (150+100 mg) vs Sitagliptin 100 mg; Pre-lunch; Time-matched change from baseline in pre-meal insulin on Day 14 was analyzed using a mixed effects model with sequence, period, treatment, the treatment by-time interaction, period-specific baseline and carryover as fixed effects. Subjects within sequences were modeled as random effects; Test type: Superiority or Other; Mean Difference (Final Values) = 1.70, 80% CI 2-sided [-1.62 to 5.01]
Statistical Analysis 10: Comparison: PF-04937319 Once-Daily (300 mg) vs Sitagliptin 100 mg; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; Mean Difference (Final Values) = 4.08, 80% CI 2-sided [0.54 to 7.62]
Statistical Analysis 11: Comparison: PF-04937319 Split-Dose (150+100 mg); Compared with Baseline (Pre-dinner); Test type: Superiority or Other; Mean Difference (Final Values) = -0.70, 80% CI 2-sided [-3.66 to 2.27]
Statistical Analysis 12: Comparison: PF-04937319 Once-Daily (300 mg); Compared with Baseline (Pre-dinner); Test type: Superiority or Other; Mean Difference (Final Values) = 5.06, 80% CI 2-sided [1.70 to 8.43]
Statistical Analysis 13: Comparison: Sitagliptin 100 mg; Compared with Baseline (Pre-dinner); Test type: Superiority or Other; Mean Difference (Final Values) = 3.42, 80% CI 2-sided [-0.10 to 6.94]
Statistical Analysis 14: Comparison: PF-04937319 Split-Dose (150+100 mg) vs Sitagliptin 100 mg; Pre-dinner; Time-matched change from baseline in pre-meal insulin on Day 14 was analyzed using a mixed effects model with sequence, period, treatment, the treatment by-time interaction, period-specific baseline and carryover as fixed effects. Subjects within sequences were modeled as random effects; Test type: Superiority or Other; Mean Difference (Final Values) = -4.12, 80% CI 2-sided [-8.42 to 0.18]
Statistical Analysis 15: Comparison: PF-04937319 Once-Daily (300 mg) vs Sitagliptin 100 mg; [analysis description as in outcome 4, analysis 14]; Test type: Superiority or Other; Mean Difference (Final Values) = 1.64, 80% CI 2-sided [-2.60 to 5.89]

5. Secondary Outcome: Incidence of All Causality Treatment-Emergent Adverse Event by Preferred Term (Frequency Rate >5%)
Time Frame: Day 1 up to Day 14
Population: The safety analysis set was all participants who received at least one dose of randomized study treatment. HAEs meeting protocol definition were summarized descriptively by treatment.
Measure: Number; unit: participants
Groups:
- Metformin Run-in: Participants were instructed to take the morning dose of the study medication and at least 1 dose of open label metformin at the same time of day with the morning meal each day.
Arm/Group | Metformin Run-in | PF-04937319 Split-Dose (150+100 mg) | PF-04937319 Once-Daily (300 mg) | Sitagliptin 100 mg
Number analyzed (Participants) | 43 | 31 | 30 | 30
participants
  Participants evaluable for AEs | 43 | 31 | 30 | 30
  Participants with AEs having a frequency rate >5% | 3 | 16 | 19 | 12
  Participants with hypoglycaemia | 2 | 11 | 14 | 4
  Participants with Headache | 0 | 4 | 4 | 4
  Participants with Back pain | 0 | 2 | 1 | 2
  Participants with Diarrhoea | 1 | 0 | 2 | 2
  Participants with Musculoskeletal pain | 0 | 1 | 2 | 1
  Participants with Pain in extremity | 0 | 1 | 2 | 1
  Participants with Cough | 0 | 1 | 0 | 2

6. Secondary Outcome: Frequency of Laboratory Test Abnormalities Reported in Any Treatment Group
Description: The total number of participants with laboratory test abnormalities (without regard to baseline abnormality) was assessed.
Time Frame: Day 1 up to Day 14
Population: The safety analysis set was all participants who received at least one dose of randomized study treatment.
Measure: Number; unit: participants
Arm/Group | PF-04937319 Split-Dose (150+100 mg) | PF-04937319 Once-Daily (300 mg) | Sitagliptin 100 mg
Number analyzed (Participants) | 31 | 30 | 27
participants
  Total neutrophils (abs) (10^3/mm^3) <0.8 × LLN | 1 | 0 | 0
  Eosinophils (abs) (10^3/mm^3) >1.2 × ULN | 0 | 0 | 1
  Triglycerides (mg/dL) >1.3 × ULN | 2 | 0 | 2
  Phosphate (mg/dL)<0.8 × LLN | 1 | 0 | 0
  Glucose (mg/dL)>1.5 × ULN | 16 | 12 | 14
  Creatine kinase (U/L) >2.0 × ULN | 1 | 1 | 0
  Urine glucose (qual) ≥1 | 8 | 4 | 5
  Urine nitrite ≥1 | 2 | 3 | 1
  Urine leukocyte esterase ≥1 | 1 | 1 | 2
  Urine WBC (/HPF) ≥20 | 1 | 1 | 1

7. Secondary Outcome: Change From Baseline in Body Weight (kg)
Time Frame: Day 1 up to Day 14
Population: The safety analysis set was all participants who received at least one dose of randomized study treatment.
Measure: Mean (Standard Error); unit: kg
Arm/Group | PF-04937319 Split-Dose (150+100 mg) | PF-04937319 Once-Daily (300 mg) | Sitagliptin 100 mg
Number analyzed (Participants) | 31 | 30 | 26
kg | 0.50 (0.313) | 0.30 (0.545) | 0.05 (0.215)
Statistical Analysis 1: Comparison: PF-04937319 Split-Dose (150+100 mg); Compared with baseline; Test type: Superiority or Other; Mean Difference (Final Values) = 0.80, 80% CI 2-sided [0.21 to 1.39]
Statistical Analysis 2: Comparison: PF-04937319 Once-Daily (300 mg); Compared with baseline; Test type: Superiority or Other; Mean Difference (Final Values) = 0.25, 80% CI 2-sided [-0.43 to 0.93]
Statistical Analysis 3: Comparison: Sitagliptin 100 mg; Compared with baseline; Test type: Superiority or Other; Mean Difference (Final Values) = -0.26, 80% CI 2-sided [-0.92 to 0.40]
Statistical Analysis 4: Comparison: PF-04937319 Split-Dose (150+100 mg) vs Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 1.06, 80% CI 2-sided [0.17 to 1.95]
Statistical Analysis 5: Comparison: PF-04937319 Once-Daily (300 mg) vs Sitagliptin 100 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.51, 80% CI 2-sided [-0.45 to 1.47]

8. Secondary Outcome: Number of Participants With Vital Signs Data Met Criteria of Potential Clinical Concern
Description: Vital signs included blood pressure (BP; supine, sitting and standing) and pulse rate. Vital signs criteria of potential clinical concern were 1), BP: sitting systolic BP (SBP) greater than or equal to (>=) 30 millimeters of mercury (mm Hg) change from baseline, sitting SBP =<20 mmHg change from baseline, supine/sitting/standing SBP less than (<) 90 mm Hg; sitting diastolic BP (DBP) >=20 mm Hg change from baseline, sitting SBP =<20 mmHg change from baseline, supine/sitting/standing DBP <50 mm Hg; 2), pulse rate (supine): <40 or greater than (>) 120 beats per minute (bpm).
Time Frame: Day 1 up to Day 14
Population: The safety analysis set was all participants who received at least one dose of randomized study treatment.
Measure: Number; unit: participants
Arm/Group | PF-04937319 Split-Dose (150+100 mg) | PF-04937319 Once-Daily (300 mg) | Sitagliptin 100 mg
Number analyzed (Participants) | 31 | 30 | 29
participants
  Sitting SBP <90 mm Hg | 0 | 0 | 0
  Sitting DBP <50 mm Hg | 0 | 0 | 1
  Sitting Pulse Rate <40 bpm | 0 | 0 | 0
  Sitting Pulse Rate >120 bpm | 0 | 0 | 0
  Increase:sitting SBP≥30 mm Hg | 1 | 1 | 2
  Increase:sitting DBP≥20 mm Hg | 0 | 1 | 0
  Decrease:sitting SBP≥30 mm Hg | 2 | 2 | 2
  Decrease:sitting DBP≥30 mm Hg | 0 | 0 | 2

9. Secondary Outcome: Number of Participants With Post-baseline Electrocardiograms (ECGs) Data Met Criteria of Potential Clinical Concern
Description: ECG criteria of potential clinical concern were 1), PR interval: >=300 milliseconds (msec); >=25% increase when baseline >200 msec; or increase >=50% when baseline <=200 msec; 2), QRS interval: >=140 msec; >=50% increase from baseline; 3), QTc interval using Fridericia's formula (QTcF interval): absolute value >=450 - <480 msec, >=480-<500 msec, >500 msec; absolute change 30 - <60, >=60 msec.
Time Frame: Day 1 up to Day 14
Population: The safety analysis set was all participants who received at least one dose of randomized study treatment.
Measure: Number; unit: participants
Arm/Group | PF-04937319 Split-Dose (150+100 mg) | PF-04937319 Once-Daily (300 mg) | Sitagliptin 100 mg
Number analyzed (Participants) | 31 | 30 | 29
participants
  PR interval >=300 msec, n=31,30,29 | 0 | 0 | 0
  QRS interval >=140 msec, n=31,30,29 | 0 | 0 | 0
  QTcF interval 450-480 msec, n=31,30,29 | 2 | 1 | 1
  QTcF interval 480-500 msec, n=31,30,29 | 0 | 0 | 0
  QTcF interval >=500 msec, n=31,30,29 | 0 | 0 | 0
  PR interval increase >=25%/50%, n=31,30,29 | 0 | 0 | 0
  QRS interval increase >=50%, n=31,30,29 | 0 | 0 | 0
  QTcF increase 30-60 msec, n=31,30,29 | 0 | 0 | 0
  QTcF increase >=60 msec, n=31,30,29 | 0 | 0 | 0

10. Secondary Outcome: Plasma PF-04937319 Area Under the Concentration Time Curve From Time 0 to 24 Hours (AUC24) of PF-04937319 at Day 14
Description: The PK parameters were summarized descriptively by treatment as appropriate. Two (2) PK parameters specified in the protocol and SAP were not reported: AUClast was not reported since it was the same as AUC24 in this study, and apparent volume of distribution (Vz/F) was not reported since the log-linear terminal phase of the concentration-time profiles was not consistently well characterized in the 24-hour sampling period.
Time Frame: Predose, 1.5, 3, 5, 6.5, 8, 11, 12.5, and 14 hours on Days 0 and 14; and predose on Days 7 and 15.
Population: The PK population was defined as all randomized participants who received at least 1 dose of PF 04937319 and who had at least 1 PK sample with reported concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | PF-04937319 Split-Dose (150+100 mg) | PF-04937319 Once-Daily (300 mg)
Number analyzed (Participants) | 31 | 30
ng•hr/mL | 10710 (43) | 11810 (47)

11. Secondary Outcome: Plasma PF-04937319 Apparent Clearance (CL/F) on Day 14
Description: The PK parameters were summarized descriptively by treatment as appropriate. Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population PK modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Predose, 1.5, 3, 5, 6.5, 8, 11, 12.5, and 14 hours on Days 0 and 14; and predose on Days 7 and 15.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | PF-04937319 Split-Dose (150+100 mg) | PF-04937319 Once-Daily (300 mg)
Number analyzed (Participants) | 31 | 30
mL/min | 389.2 (43) | 423.3 (47)

12. Secondary Outcome: Plasma PF-04937319 Average Concentration Over the 24-hour Period (Cav) on Day 14
Description: Cav was average concentration over the 24-hour period. The PK parameters were summarized descriptively by treatment as appropriate.
Time Frame: Predose, 1.5, 3, 5, 6.5, 8, 11, 12.5, and 14 hours on Days 0 and 14; and predose on Days 7 and 15.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04937319 Split-Dose (150+100 mg) | PF-04937319 Once-Daily (300 mg)
Number analyzed (Participants) | 31 | 30
ng/mL | 446.1 (43) | 492.0 (47)

13. Secondary Outcome: Plasma PF-04937319 Highest Observed Concentration (Cmax) on Day 14
Description: Cmax was highest observed concentration. The PK parameters were summarized descriptively by treatment as appropriate.
Time Frame: Predose, 1.5, 3, 5, 6.5, 8, 11, 12.5, and 14 hours on Days 0 and 14; and predose on Days 7 and 15.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04937319 Split-Dose (150+100 mg) | PF-04937319 Once-Daily (300 mg)
Number analyzed (Participants) | 31 | 30
ng/mL | 776.6 (39) | 980.5 (38)

14. Secondary Outcome: Plasma PF-04937319 Lowest Observed Concentration During the 24-hour Period (Cmin) on Day 14
Description: Cmin lowest observed concentration during the 24-hour period. The PK parameters were summarized descriptively by treatment as appropriate.
Time Frame: Predose, 1.5, 3, 5, 6.5, 8, 11, 12.5, and 14 hours on Days 0 and 14; and predose on Days 7 and 15.
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04937319 Split-Dose (150+100 mg) | PF-04937319 Once-Daily (300 mg)
Number analyzed (Participants) | 31 | 30
ng/mL | 101.9 (602) | 131.0 (265)

15. Secondary Outcome: Plasma PF-04937319 Time for Cmax (Tmax) on Day 14
Description: Tmax was time of maximum concentration. The PK parameters were summarized descriptively by treatment as appropriate.
Time Frame: Predose, 1.5, 3, 5, 6.5, 8, 11, 12.5, and 14 hours on Days 0 and 14; and predose on Days 7 and 15.
Population: as for outcome 10
Measure: Median (Full Range); unit: hour
Arm/Group | PF-04937319 Split-Dose (150+100 mg) | PF-04937319 Once-Daily (300 mg)
Number analyzed (Participants) | 31 | 30
hour | 6.50 (602) [3.00 to 11.0] | 5.00 (265) [1.50 to 12.5]

ADVERSE EVENTS:
Groups:
- Metformin Run-in: Sponsor-provided, open-label metformin was administered from the run-in visit to the follow-up visit, inclusive, and it was provided as 500 mg immediate-release tablets.
- PF-04937319 150+100 mg (Split Dose): Participants were instructed to take the morning dose of PF-04937319 150 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day. In addition, the second dose of the study medication (PF-04937319 100 mg) should have been taken with the lunch meal approximately 5±1 hours after the morning dose, each day, for 14±2 days.
- PF-04937319 300 mg (Once Daily): Participants were instructed to take the morning dose of PF-04937319 300 mg and at least 1 dose of open label metformin at the same time of day with the morning meal each day. In addition, the second dose of the study medication (placebo) should have been taken with the lunch meal approximately 5±1 hours after the morning dose, each day, for 14±2 days.
Arm/Group | Metformin Run-in | PF-04937319 150+100 mg (Split Dose) | PF-04937319 300 mg (Once Daily) | Sitagliptin 100 mg
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/31 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 3/43 | 16/31 | 19/30 | 12/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin Run-in (N=43) | PF-04937319 150+100 mg (Split Dose) (N=31) | PF-04937319 300 mg (Once Daily) (N=30) | Sitagliptin 100 mg (N=30)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 11 | 14 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1
Headache (Nervous system disorders) | 0 | 4 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.